CLINICAL TRIAL: NCT01956123
Title: A Controlled, Assessor-blind, Parallel Groups, Multicentre, Multinational Trial Evaluating the Immunogenicity of FE 999049 in Repeated Cycles of Controlled Ovarian Stimulation in Women Undergoing an Assisted Reproductive Technology Programme
Brief Title: Evidence-based Stimulation Trial With Human rFSH in Europe and Rest of World 2
Acronym: ESTHER-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000071; 2013-001616-30 (EudraCT Number); U1111-1147-6922 (Other: WHO)
Record Dates: First submitted 2013-08-16; First posted 2013-10-08 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2018-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta; FE 999049; follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Follitropin Delta (FE 999049) (COS cycle 2)
  Interventions: Drug: Follitropin Delta (FE 999049)
- B (Active Comparator): Follitropin Alfa (GONAL-F) (COS cycle 2)
  Interventions: Drug: Follitropin Alfa (GONAL-F)
- C (Experimental): Follitropin Delta (FE 999049) (COS cycle 3)
  Interventions: Drug: Follitropin Delta (FE 999049)
- D (Active Comparator): Follitropin Alfa (GONAL-F) (COS cycle 3)
  Interventions: Drug: Follitropin Alfa (GONAL-F)

INTERVENTIONS:
Drug: Follitropin Delta (FE 999049)
  Arms: A; C
Drug: Follitropin Alfa (GONAL-F)
  Arms: B; D

SUMMARY:
This trial investigates the immunogenicity of FE 999049 in repeated cycles.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Documents signed prior to screening evaluations related to this protocol
* Participation in the pivotal efficacy trial (trial 000004/ESTHER-1)
* Anti-FSH antibody results from baseline and at least one post-dosing assessment in the previous cycle(s) available.
* Having undergone the oocyte retrieval procedure, or having had cycle cancellation prior to oocyte retrieval due to poor ovarian response or excessive ovarian response, in the previous cycle(s).
* Failure to achieve ongoing pregnancy in the previous cycle(s).

Exclusion Criteria:

* Non-compliance to protocol compliance in the previous cycle(s).
* Having undergone any stimulation with gonadotropins since the end-of-trial / end-of-cycle visit in the previous cycle
* One or more follicles ≥10 mm observed on the transvaginal ultrasound prior to start of dosing on stimulation day 1
* Severe OHSS in a previous cycle.
* Any clinically relevant change to any of the eligibility criteria in the previous cycle(s).
* Clinically relevant medical history since the previous cycle which precludes gonadotropin stimulation or is associated with a reduced chance of pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 513 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (13):
- UZ Brussel (there may be other sites in this country), Brussels, Belgium
- Fertilitat and PUC-RS (there may be other sites in this country), Porto Alegre, Brazil
- Canada (3):
  - Pacific Centre for Reproductive Medicine, Burnaby, British Columbia
  - Olive Fertility Centre, Vancouver, British Columbia
  - Ottawa Fertility Centre, Ottawa, Ontario
- IVF CUBE SE (there may be other sites in this country), Prague, Czechia
- Rigshospitalet Fertilitetsklinikken (there may be other sites in this country), Copenhagen, Denmark
- Department of Endocrine Gynaecology and Reproductive Medicine, Hôpital Jeanne de Flandre (there may be other sites in this country), Lille, France
- Centro Natalità San Raffaele (there may be other sites in this country), Milan, Italy
- The nOvum Clinic (there may be other sites in this country), Warsaw, Poland
- IVF & Reproductive Genetics Center (there may be other sites in this country), Moscow, Russia
- IVI Sevilla (there may be other sites in this country), Seville, Spain
- Glasgow Centre for Reproductive Medicine Ltd. (there may be other sites in this country), Glasgow, United Kingdom

REFERENCES:
- [Result] Havelock J, Aaris Henningsen AK, Mannaerts B, Arce JC; ESTHER-1 and ESTHER-2 Trial Groups. Pregnancy and neonatal outcomes in fresh and frozen cycles using blastocysts derived from ovarian stimulation with follitropin delta. J Assist Reprod Genet. 2021 Oct;38(10):2651-2661. doi: 10.1007/s10815-021-02271-5. Epub 2021 Jul 13. PMID 34254211
- [Result] Fernandez-Sanchez M, Fatemi H, Garcia-Velasco JA, Heiser PW, Daftary GS, Mannaerts B. Incidence and severity of ovarian hyperstimulation syndrome (OHSS) in high responders after gonadotropin-releasing hormone (GnRH) agonist trigger in "freeze-all" approach. Gynecol Endocrinol. 2023 Dec;39(1):2205952. doi: 10.1080/09513590.2023.2205952. PMID 37156263
- [Derived] Nelson SM, Larsson P, Mannaerts BMJL, Nyboe Andersen A, Fauser BCJM. Anti-Mullerian hormone variability and its implications for the number of oocytes retrieved following individualized dosing with follitropin delta. Clin Endocrinol (Oxf). 2019 May;90(5):719-726. doi: 10.1111/cen.13956. Epub 2019 Mar 18. PMID 30801744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 investigational sites included participants to the trial : 3 in Belgium, 3 in Brazil, 3 in Canada, 3 in the Czech Republic, 2 in Denmark, 2 in Italy, 2 in Poland, 2 in Russia, 10 in Spain and 2 in United Kingdom.
Pre-assignment Details: Participants who participated in Trial 000004 (NCT01956110) (controlled ovarian stimulation [COS] cycle 1) & failed to achieve ongoing pregnancy were eligible for the trial. For COS cycle 2, 520 participants were screened and 513 enrolled. For COS cycle 3, 190 participants were screened and 189 enrolled. Participants were exposed to the same IMP as in COS cycle 1.
Groups:
- FE 999049 (COS Cycle 2): FE 999049 was administered as single daily subcutaneous injections in the abdomen. The dose was determined based on the ovarian response in COS cycle 1. The daily FE 999049 dose was fixed throughout the stimulation period and maximum allowed daily dose was 18 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- GONAL-F (COS Cycle 2): Follitropin Alfa (GONAL-F) was administered as single daily subcutaneous injections in the abdomen. The starting dose was determined based on the ovarian response in COS cycle 1. The GONAL-F starting dose was fixed for the first 5 days after which it could be adjusted by 75 international units (IU) based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- FE 999049 (COS Cycle 3): FE 999049 was administered as single daily subcutaneous injections in the abdomen. The dose was determined based on the ovarian response in COS cycle 2. The daily FE 999049 dose was fixed throughout the stimulation period and maximum allowed daily dose was 24 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- GONAL-F (COS Cycle 3): GONAL-F was administered as single daily subcutaneous injections in the abdomen. The starting dose was determined based on the ovarian response in COS cycle 2. The GONAL-F starting dose was fixed for the first 5 days after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
Period: COS Cycle 2
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Started | 252 | 261 | 0 | 0
Completed | 238 | 254 | 0 | 0
Not Completed | 14 | 7 | 0 | 0
Not completed — Protocol Violation | 8 | 3 | 0 | 0
Not completed — Adverse Event | 3 | 4 | 0 | 0
Not completed — Personal Reasons | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: COS Cycle 3
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Started | 0 | 0 | 95 (Participants in COS cycle 2 who failed to achieve an ongoing pregnancy could undergo COS cycle 3) | 93 (Participants in COS cycle 2 who failed to achieve an ongoing pregnancy could undergo COS cycle 3)
Completed | 0 | 0 | 89 | 91
Not Completed | 0 | 0 | 6 | 2
Not completed — Protocol Violation | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 0
Not completed — Personal Reasons | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GONAL-F (COS Cycle 2): GONAL-F was administered as single daily subcutaneous injections in the abdomen. The starting dose was determined based on the ovarian response in COS cycle 1. The GONAL-F starting dose was fixed for the first 5 days after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- Total: Total of all reporting groups
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | Total
Number analyzed (Participants) | 252 | 261 | 513
Age, Categorical [Count of Participants; unit: Participants] — Population: Only participants who participated in COS cycle 2 but failed to achieve an ongoing pregnancy could undergo COS cycle 3.
  Participants
    COS cycle 2: <=18 years | 0 | 0 | 0
    COS cycle 2: Between 18 and 65 years | 252 | 261 | 513
    COS cycle 2: >=65 years | 0 | 0 | 0
    COS cycle 3: number analyzed (Participants) | 95 | 93 | 188
    COS cycle 3: <=18 years | 0 | 0 | 0
    COS cycle 3: Between 18 and 65 years | 95 | 93 | 188
    COS cycle 3: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only participants who participated in COS cycle 2 but failed to achieve an ongoing pregnancy could undergo COS cycle 3.
  Participants
    COS cycle 2: Female | 252 | 261 | 513
    COS cycle 2: Male | 0 | 0 | 0
    COS cycle 3: number analyzed (Participants) | 95 | 93 | 188
    COS cycle 3: Female | 95 | 93 | 188
    COS cycle 3: Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion (Percentage) of Subjects With Treatment-induced Anti-Follicle-Stimulating Hormone (FSH) Antibodies After up to Two Repeated Controlled Ovarian Stimulation Cycles
Description: The proportion (percentage) of participants with at least one treatment-induced anti-FSH antibody response at any time point is presented. The cumulative incidences in COS cycle 2 and COS cycle 3 divided by participants in COS cycle 2 are presented. Participants with observations in both cycles are only counted once.
Time Frame: Stimulation day 1, 7-10 days after last FE 999049 or GONAL-F dose and 21-28 days after last FE 999049 or GONAL-F dose
Population: Safety analysis set (all exposed participants).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2)
Number analyzed (Participants) | 252 | 261
Percentage of participants | 0.79 [0.10 to 2.84] | 0.38 [0.01 to 2.12]

2. Secondary Outcome: Proportion (Percentage) of Subjects With Treatment-induced Anti-FSH Antibodies With Neutralising Capacity After up to Two Repeated Controlled Ovarian Stimulation Cycles
Description: The proportion (percentage) of participants with treatment-induced anti-FSH antibodies with neutralising capacity at any time point is presented. The cumulative incidences in COS cycle 2 and COS cycle 3 divided by participants in COS cycle 2 are presented. Participants with observations in both cycles are only counted once.
Time Frame: Stimulation day 1, 7-10 days after last FE 999049 or GONAL-F dose and 21-28 days after last FE 999049 or GONAL-F dose
Population: Safety analysis set (all exposed participants).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2)
Number analyzed (Participants) | 252 | 261
Percentage of participants | 0.00 [0.00 to 1.45] | 0.00 [0.00 to 1.40]

3. Secondary Outcome: Proportion (Percentage) of Subjects With Treatment-induced Anti-FSH Antibodies, Overall as Well as With Neutralising Capacity, After One and After Two Repeated Controlled Ovarian Stimulation Cycles
Description: The proportion (percentage) of participants with treatment-induced anti-FSH antibodies, overall as well as with neutralising capacity, after one and after two repeated COS cycles is presented.
Time Frame: Stimulation day 1, 7-10 days after last FE 999049 or GONAL-F dose and 21-28 days after last FE 999049 or GONAL-F dose
Population: Safety analysis set (all exposed participants).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants
  Treatment-induced anti-FSH antibodies | 0.79 [0.10 to 2.84] | 0.38 [0.01 to 2.12] | 1.05 [0.03 to 5.73] | 1.08 [0.03 to 5.85]
  Antibodies with neutralising capacity | 0.00 [0.00 to 1.45] | 0.00 [0.00 to 1.40] | 0.00 [0.00 to 3.81] | 0.00 [0.00 to 3.89]

4. Secondary Outcome: Proportion (Percentage) of Subjects With Early Ovarian Hyperstimulation Syndrome (OHSS) (Including OHSS of Moderate/Severe Grade) and/or Preventive Interventions for Early OHSS for Each Controlled Ovarian Stimulation Cycle
Description: The proportion (percentage) of participants with early OHSS, early OHSS of moderate or severe grade, preventive interventions for early OHSS, early OHSS and/or preventive interventions for early OHSS, and early OHSS of moderate or severe grade and/or preventive interventions for early OHSS are presented.
Time Frame: ≤9 days after triggering of final follicular maturation.
Population: Modified intention-to-treat (mITT) analysis set (all exposed participants). This is equivalent to the full analysis set (FAS).
Measure: Number; unit: Percentage of participants
Groups:
- GONAL-F (COS Cycle 2): Follitropin Alfa (GONAL-F) was administered as single daily subcutaneous injections in the abdomen. The starting dose was determined based on the ovarian response in COS cycle 1. The GONAL-F starting dose was fixed for the first 5 days after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants
  Early OHSS (any grade) | 0.8 | 2.3 | 1.1 | 0.0
  Early OHSS (moderate/severe) | 0.0 | 1.9 | 0.0 | 0.0
  Any preventive intervention | 1.6 | 1.9 | 0.0 | 1.1
  Early OHSS (any grade) / preventive | 2.0 | 3.8 | 1.1 | 1.1
  Early OHSS (moderate/severe) / preventive | 1.6 | 3.8 | 0.0 | 1.1

5. Secondary Outcome: Proportion (Percentage) of Subject With Cycle Cancellation Due to Poor Ovarian Response or Excessive Ovarian Response for Each Controlled Ovarian Stimulation Cycle
Description: Proportion (percentage) of participants with cycle cancellation due to poor ovarian response, excessive ovarian response, and triggering with gonadotropin-releasing hormone (GnRH) agonist are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: mITT analysis set (all exposed participants). This is equivalent to the FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants
  Cycle cancelled due to poor ovarian response | 2.0 | 3.8 | 2.1 | 2.2
  Cycle cancelled due to excessive ovarian response | 0.4 | 0.0 | 0.0 | 0.0
  Triggering with GnRH agonist | 0.4 | 0.8 | 0.0 | 1.1

6. Secondary Outcome: Vital Pregnancy Rate for Each Controlled Ovarian Stimulation Cycle
Description: Vital pregnancy was defined as at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after blastocyst transfer.
Time Frame: 5-6 weeks after blastocyst transfer
Population: mITT analysis set (all exposed participants). This is equivalent to the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants | 29.4 [23.8 to 35.4] | 27.2 [21.9 to 33.0] | 27.4 [18.7 to 37.5] | 29.0 [20.1 to 39.4]

7. Secondary Outcome: Implantation Rate for Each Controlled Ovarian Stimulation Cycle
Description: Implantation rate was defined as the number of gestational sacs 5-6 weeks after transfer divided by number of blastocysts transferred.
Time Frame: 5-6 weeks after blastocyst transfer
Population: Participants with blastocyst transfer. In COS cycle 2, a total of 254 and 271 blastocysts were transferred in the FE 999049 and GONAL-F groups, respectively. In COS cycle 3, a total of 132 and 121 blastocysts were transferred in the FE 999049 and GONAL-F groups, respectively.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 211 | 221 | 82 | 75
Percentage | 34.6 [28.8 to 40.8] | 30.6 [25.2 to 36.5] | 28.8 [21.2 to 37.3] | 32.2 [24.0 to 41.3]

8. Secondary Outcome: Ongoing Pregnancy Rate for Each Controlled Ovarian Stimulation Cycle
Description: Ongoing pregnancy rate was defined as at least one intrauterine viable fetus 10-11 weeks after blastocyst transfer.
Time Frame: 10-11 weeks after blastocyst transfer
Population: mITT analysis set (all exposed participants). This is equivalent to FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants | 27.8 [22.3 to 33.7] | 25.7 [20.5 to 31.4] | 27.4 [18.7 to 37.5] | 28 [19.1 to 38.2]

9. Secondary Outcome: Ongoing Implantation Rate for Each Controlled Ovarian Stimulation Cycle
Description: Ongoing implantation rate was defined as the number of intrauterine viable fetuses 10-11 weeks after transfer divided by number of blastocysts transferred.
Time Frame: 10-11 weeks after blastocyst transfer
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 211 | 221 | 82 | 75
Percentage | 28.7 [23.3 to 34.7] | 25.5 [20.4 to 31.1] | 25.0 [17.9 to 33.3] | 28.9 [21.0 to 37.9]

10. Secondary Outcome: Frequency of Injection Site Reactions (Redness, Pain, Itching, Swelling and Bruising) Assessed by the Subject During the Stimulation Period for Each Controlled Ovarian Stimulation Cycle
Description: Participants self-assessed injection site reactions (redness, itching, pain, swelling and bruising) immediately, 30 minutes and 24 hours after each injection. The injection site reactions were assessed as none, mild, moderate and severe. The frequency of injection site reactions (mild, moderate or severe) based on all assessment performed is presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: Safety analysis set (all exposed participants).
Measure: Number; unit: Percentage of events
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of events | 3.0 | 2.4 | 2.8 | 2.3

11. Secondary Outcome: Proportion (Percentage) of Subjects With Late OHSS (Including OHSS of Moderate/Severe Grade) for Each Controlled Ovarian Stimulation Cycle
Description: Late OHSS was defined as OHSS with onset >9 days after triggering of final follicular maturation.
Time Frame: >9 days after triggering of final follicular maturation
Population: Safety analysis set (all exposed participants).
Measure: Number; unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants
  Late OHSS (any grade) | 0.4 | 0.8 | 1.1 | 1.1
  Late OHSS (moderate/severe) | 0.0 | 0.8 | 0.0 | 1.1

12. Secondary Outcome: Technical Malfunctions of the Administration Pen for Each Controlled Ovarian Stimulation Cycle
Description: Incidences of confirmed technical malfunction of administration pen are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: Safety analysis set (all exposed participants).
Measure: Number; unit: Percentage of participants
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
Number analyzed (Participants) | 252 | 261 | 95 | 93
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from signed informed consent to the end-of-cycle visit for COS cycle 2 (up to approximately 4.5 months) and again from screening to the end-of-cycle visit for COS cycle 3 (up to approximately 4.5 months).
Description: AEs with onset after start of first administration of IMP and before the end-of-cycle were considered treatment-emergent and are presented for the safety analysis set.
Arm/Group | FE 999049 (COS Cycle 2) | GONAL-F (COS Cycle 2) | FE 999049 (COS Cycle 3) | GONAL-F (COS Cycle 3)
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/261 | 0/95 | 0/93
Serious Adverse Events (participants affected / at risk) | 4/252 | 4/261 | 0/95 | 1/93
Other Adverse Events (participants affected / at risk) | 70/252 | 77/261 | 26/95 | 34/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (COS Cycle 2) (N=252) | GONAL-F (COS Cycle 2) (N=261) | FE 999049 (COS Cycle 3) (N=95) | GONAL-F (COS Cycle 3) (N=93)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (COS Cycle 2) (N=252) | GONAL-F (COS Cycle 2) (N=261) | FE 999049 (COS Cycle 3) (N=95) | GONAL-F (COS Cycle 3) (N=93)
Procedural pain (Injury, poisoning and procedural complications) | 13 (14) | 17 (20) | 5 (6) | 8 (8)
Headache (Nervous system disorders) | 19 (24) | 27 (34) | 11 (12) | 13 (15)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 8 (8) | 9 (9) | 4 (4)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 13 (15) | 10 (11) | 3 (3) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 9 (9) | 5 (5) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 14 (14) | 11 (12) | 3 (3) | 5 (5)
Pelvic discomfort (Reproductive system and breast disorders) | 6 (6) | 13 (14) | 0 (0) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.